CLINICAL TRIAL: NCT03446105
Title: Promoting Quality of Life Among Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Carla Berg, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00086979
Record Dates: First submitted 2018-02-21; First posted 2018-02-26 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Cancer
Keywords: Cancer survivor; App-based intervention; Behavioral intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned (stratified by age and sex) to one of the treatment conditions in a 2:1 ratio (2 to intervention: 1 to attention control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App-based behavioral intervention (Experimental): Participants randomized to this study arm will take part in the Achieving Wellness After Kancer in Early life (AWAKE) behavioral intervention for 8 weeks.
  Interventions: Behavioral: App-based behavioral intervention
- Attention control group (Active Comparator): Participants randomized to this study arm will take part in a behavioral intervention and coaching for 8 weeks.
  Interventions: Behavioral: Attention control group

INTERVENTIONS:
Behavioral: App-based behavioral intervention — Achieving Wellness After Kancer in Early life (AWAKE) is a behavioral intervention that includes a smartphone app and coaching. AWAKE contains eight modules, and participants will complete the one module every week. App functioning will facilitate weekly homework assignments and include health education messaging, the ability to track progress toward goals over time via self-monitoring and graphical depictions of progress, audio-recordings of guided imagery exercises and relaxation exercises (e.g., progressive muscle relaxation), videos of topic-related inspirational material, and a portal for interacting with the coach. The coach will call each intervention participant weekly. Each coaching session will last roughly 30 minutes and involve four segments that will correspond to the module for the week. The coach will send daily text messages to participants encouraging their goal pursuits and providing other sources of support related to that week's homework.
  Other Names: AWAKE
  Arms: App-based behavioral intervention
Behavioral: Attention control group — The attention control group will receive the same components as the intervention group, but the educational modules will contain different content than those receiving the AWAKE intervention.
  Arms: Attention control group

SUMMARY:
This study expands on a prior pilot study to refine the intervention messaging to focus on goal-oriented thinking, include a coach, and extend the intervention to a larger sample of young adult cancer survivors (aged 18-39 years) recruited from two National Cancer Institute (NCI)-designated cancer centers (Emory's Winship Cancer Institute in Atlanta; University of Kentucky's Markey Cancer Center in Lexington). Participants will be randomly assigned (stratified by age and sex) to one of the 8-week treatment conditions in a 2:1 ratio (2 to intervention: 1 to attention control).

DETAILED DESCRIPTION:
Young adulthood is a critical time for negotiating several life transitions and establishing and pursuing important life goals. Unfortunately, a cancer diagnosis disrupts this period of life for more than 60,000 people annually in the U.S. Compared to those without a history of cancer, young adult cancer survivors report poorer mental and physical health; moreover, they report significantly greater disruption in their goal pursuits than cancer survivors diagnosed at a later age. However, this high-risk group has been underserved and understudied, particularly in terms of intervention research to address these sequelae. Hope, a positive psychology construct that taps the ways in which people choose and pursue goals, is particularly relevant to this population. Additionally, higher hope is related to engaging in health promoting behaviors and living healthier lifestyles, which reduces risk of disease and adverse late effects and ultimately increase quality of life (QOL). The research team has pioneered a app-based behavioral intervention called Achieving Wellness After Kancer in Early life (AWAKE), aimed at promoting healthy lifestyles - specifically targeting mental health and positive health behaviors - among young adult cancer survivors. The proposed study will refine the intervention messaging to focus on goal-oriented thinking, include a coach, and extend the prior pilot work to a larger sample of young adult cancer survivors (aged 18-39 years) recruited from two NCI-designated cancer centers (Emory's Winship Cancer Institute in Atlanta; University of Kentucky's Markey Cancer Center in Lexington). In this randomized controlled trial, recipients of the AWAKE intervention will be compared to an attention control group.

The specific aims of this study are to:

Aim 1. Test the feasibility and acceptability of AWAKE among intervention participants. The primary feasibility indicators are participation rates and retention rates. The primary acceptability indicators are use of and satisfaction with intervention components.

Aim 2. Estimate effect sizes of AWAKE vs. control at 2 and 6 months to inform sample size calculations for the subsequent efficacy trial. The primary outcome is changes in hope, per the Trait Hope Scale. The secondary outcome is changes in quality of life, per the 36-Item Short Form Health Survey (SF-36) and the Functional Assessment of Cancer Therapy - General (FACT-G).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 39, as of January 15th, 2017
* Speak English
* Be within two years of cancer treatment completion (since January 15th, 2015)
* Have a functioning smartphone and reliable internet access
* Be willing to complete study activities

Exclusion Criteria:

* Cancer recurrence since treatment completion
* Diagnosis of a central nervous system cancer (to ensure requisite mental/emotional functioning to engage in the program)
* Diagnosis of a thyroid cancer
* History of alcohol or drug dependency in the past year, or psychosis, bipolar disorder, or major depressive disorder
* In hospice

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Adult Trait Hope Scale Score | Baseline, Month 2, Month 6
  The Adult Trait Hope Scale is a 12-item survey where respondents indicate how true a statement is on a scale of 1 (definitely false) to 8 (definitely true). The Hope Scale includes two subscales of four items each plus four distracter items. Higher scores on the Pathways subscale (example question: "I can think of many ways to get out of a jam") indicate higher levels of pathways thinking. Higher scores on the Agency subscale (example question: "I energetically pursue my goals") indicate higher levels of agency thinking. The subscales will be summed to obtain a total hope score. Total scores can range from 8 to 64 with higher scores indicating higher levels of hope.

SECONDARY OUTCOMES:
Change in 36-Item Short Form Health Survey (SF-36) Score | Baseline, Month 2, Month 6
  The 36-Item Short-Form Health Survey (SF-36) asks respondents to rate their health and abilities to do their usual tasks. The SF-36 uses a variety of questions and response options and includes 8 subscales (physical functioning, role limitations due to physical health, role limitations due to emotional health, energy/fatigue, emotional well-being, social functioning, pain, and general health). Responses are coded on a scale of 0 to 100 where 0 is the worst possible health and 100 is the most favorable health score. The coded responses will be summed and averaged to obtain a mean score for the entire survey.
  The SF-36 is standardized to the general population with a mean of 50 and a standard deviation of 10. Scores above 50 indicate better than average health while scores below 50 are worse than average health scores.
Change in Functional Assessment of Cancer Therapy - General (FACT-G) Score | Baseline, Month 2, Month 6
  The FACT-G is a 27-item quality of life (QOL) measure specific to cancer patients to provide insight into cancer specific factors in four dimensions (physical, social/family, emotional, functional well-being). Participants respond to a list of statements that tend to impact people with cancer by indicating how much they are impacted on a scale of 0 (not at all) to 4 (very much). Scores for negatively worded statements are reversed so that higher scores indicate positive health. Scores from the four dimensions can be summed to create a total score. Total possible scores range from 0 to 108, with higher scores indicating increased well being.

OTHER OUTCOMES:
Participation rate | Baseline
  The participation rate will be recorded to assess feasibility of the intervention.
Retention rate | Month 2, Month 6
  The retention rate will be recorded to assess feasibility of the intervention.
Use of AWAKE | Month 2
  Acceptability will be assessed by evaluating the number of participants in the intervention who use the AWAKE app. Participants will be asked about use of specific components of the app, such as watching the videos, recording health behaviors and mood, and completing homework.
Satisfaction with AWAKE | Month 2
  Participants randomized to AWAKE will receive a survey to assess their satisfaction with the intervention. Participants will indicate the usefulness of the different components of the AWAKE program as well as overall satisfaction with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Berg, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Markey Cancer Center, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: Undecided